CLINICAL TRIAL: NCT05989607
Title: Kids Rehydration During Exercise (ROAR East)
Brief Title: Kids Rehydration During Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Collaborators: Kraft Heinz Company (Industry); Arizona State University (Other)
Responsible Party: Principal Investigator, Colleen Munoz, PhD, Associate Professor, Hydration Health Center Director, University of Hartford
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 23-03-190
Record Dates: First submitted 2023-07-11; First posted 2023-08-14 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Dehydration in Children; Dehydration Following Exertion (Disorder)

STUDY DESIGN:
Intervention Model Description: randomized, counter-balanced, cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Sugar Flavored Water (Experimental): A commercially available low sugar flavored water (2.88kcal/100ml; 0.57(sugar) +0.03 (stevia)=0.60g/100ml; sodium 7.9mg/100ml).
  Interventions: Other: Lower sugar flavored water
- Plain Water (Active Comparator): Plain water (bottled, spring).
  Interventions: Other: Plain Water

INTERVENTIONS:
Other: Lower sugar flavored water — A commercially available low sugar flavored water (2.88kcal/100ml; 0.57(sugar) +0.03 (stevia)=0.60g/100ml; sodium 7.9mg/100ml).
  Arms: Low Sugar Flavored Water
Other: Plain Water — Commercially available bottled, spring water.
  Arms: Plain Water

SUMMARY:
The present study aims to measure the impact of consuming a lower sugar flavored water compared to an equal amount of plain water during exercise on selected rehydration markers in healthy children. Participants will complete two experimental visits designed to examine the differentiating effects of one of two selected beverages (1) lower sugar flavored water beverage and 2) plain water) on certain hydration markers and related perceptual variables during repeated bouts of exercise in a warm environment to induce mild dehydration.

DETAILED DESCRIPTION:
Parents of adolescent children have demonstrated a preference to remove added and larger boluses of sugar from their child's diet in accordance with accumulating health concerns. While forms of sugar are often included in oral rehydration solutions, evidence demonstrates that electrolytes such as sodium are the predominant beverage ingredients contributing to rehydration. Determining the efficacy and preference when thirsty of a flavored water beverage (with lower sugar content), compared to plain water could guide future beverage selection to achieve rehydration in young people.

Protocol:

This is a randomized, counter-balanced, cross-over design study. Thirty participants will be voluntarily enrolled (defined as the completion of assent and successful screening). Upon enrollment, participants will be familiarized to the study procedures: exercise, dietary consumption, urine sample collection, body weight measurement, bioelectrical impedance spectroscopy (BIS) analysis, and perceptual questionnaire completion. Participants will be scheduled to complete two experimental visits within three weeks of one another. Each experimental visit is designed to examine the differentiating effects of one of two selected beverages (1) lower sugar flavored water beverage and 2) plain water) on certain hydration markers and related perceptual variables during repeated bouts of exercise.

Day Before study:

Participants will consume a standardized frozen dinner (provided by the researchers) and consume at least 250 ml (8oz) of water after dinner. Food and beverages other than water will be prohibited following dinner.

Study Day:

Participants will arrive at each study visit fasted (no food or beverages within the previous eight hours, except 250 ml of plain water two to three hours prior to the experimental visit). In the event that the participant did not fast, their visit will be rescheduled. Only one visit reschedule will be offered throughout the course of their participation. Upon arrival, participants will then consume a standardized breakfast. Following breakfast (approximately 15min following completion) they will provide a urine sample, the investigators will record body weight and measure body fluids by BIS (in a prone position), and they will complete questionnaires (with appropriate guidance and in visual analogue scale format) about mouth dryness, taste pleasantness, stomach fullness, and thirst. All body weight measurements will be taken with as minimal clothing as possible; only the participant's parent/guardian will be with the participant for this measurement to protect privacy. Each participant will wear the same amount of clothing for every body weight measurement during their individual participation.

Subsequently, the participant will enter a warm room with a controlled/recorded temperature between 28-30°C (80-85°F). Then the participant will undergo a 3 hour intermittent walk, cycle, rest protocol. During the 3-h period, each participant will complete the following one hour test, three sequential times:

* 10 min walking on the treadmill at 70% of age-predicted max heart rate (~140 bpm)
* 5 min rest
* 10 min cycling on the cycle ergometer at 70 of age-predicted max heart rate (~140 bpm)
* 35 min rest

During the 3-h period, participants will be provided with the fluid volume equating to 2% of body mass losses (as determined by ongoing individual body weight difference measurements) during each one hour test (water or a lower sugar flavored water beverage); anticipated as ~200ml). During this time body weight, and urine samples, BIS, and perceptual data via questionnaires will be collected (prior to and following each exercise bout).

ELIGIBILITY:
Inclusion Criteria:

* Girls and boys age 8 to 10y
* Willing and able to walk and cycle at a moderate intensity for sequential brief exercise periods (separated by a brief rest period) repeatedly (3x) in a warm environment (80-85°F)
* Body weight ≤85th percentile for their age group

Exclusion Criteria:

* History of conditions or current use of medications known to alter body water balance (diabetes, renal disease, SSRI's, etc.)
* Current or recent (past two weeks) illness involving fever, diarrhea, and/or GI discomfort
* Physical or mental disabilities and injuries that would prevent participation in moderate-intensity treadmill walking/jogging and cycling
* Previous diagnosis of heat stroke
* Body weight ≥86th percentile for their age group

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Net fluid balance (according to body weight change) from baseline to 3 hours post exercise | baseline to 3 hours post exercise
  Net fluid balance (according to body weight change) attributable to sweat/body water losses/additions by control of food/beverage intake and urine/fecal output; post 3 hour post exercise body weight (180min) - baseline body weight (0 minutes) = net fluid balance.

SECONDARY OUTCOMES:
Hydration status change (according to urine concentration) from baseline to 3 hours post exercise | baseline to 3 hours post exercise
  Hydration status change according to urine concentration measurement (osmolality, specific gravity, and color); 3 hour post-exercise urine concentration (180min) - baseline urine concentration (0 minutes) = hydration status change.
Total and compartmental body water change (according to bioelectrical impedance spectroscopy) from baseline to 3 hours post-exercise | baseline to 3 hours post exercise
  Total and compartmental body water change (according to bioelectrical impedance spectroscopy); 3 hour post exercise kilohertz (180 minutes) - baseline kilohertz (0 minutes) = total and compartmental body water change.
Hydration-related perceptual variable change (thirst, mouth dryness, taste pleasantness) from baseline to 3 hours post-exercise | baseline to 3 hours post exercise
  Hydration-related perceptual variable change (thirst, mouth dryness, taste pleasantness; via visual analog scale, measured in millimeters, where higher millimeters represents greater perception of that variable); 3 hours post-exercise millimeters (180min) - baseline millimeters (0min) = hydration-related perceptual variable change

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Munoz, PhD, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No